CLINICAL TRIAL: NCT06341881
Title: Understanding the Need and Feasibility of Transitional Care Training Program Among Family Caregivers of Geriatric Stroke Survivors in Pakistan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber Medical University Peshawar (Other)
Responsible Party: Principal Investigator, Dr. Najma Naz, Associate Professor, Khyber Medical University Peshawar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KMU/DIR/CTU/2024/006; KMU-CTU-2024-2001 (Other: Khyber Medical University Clinical Trial Unit)
Record Dates: First submitted 2024-03-18; First posted 2024-04-02 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Stroke; Stroke, Ischemic; Stroke Hemorrhagic
Keywords: Stroke; Geriatrics; Family caregivers; Needs assessment; Nursing; Home care
MeSH Terms: conditions — Stroke; Ischemic Stroke; Hemorrhagic Stroke

STUDY DESIGN:
Intervention Model Description: The most commonly two armed parallel study design would be used to conduct the current study. The study participants in an intervention group would be compared with that of a control group. Equal number of Participants would be allocated with random assignment in the two groups.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The study participants would not be informed of what group they are in. Independent outcome assessors would be utilized for the assessment. Further outcomes assessors and data analysts' would be kept unaware of intervention or group allocations to carry out their assessment after inclusion of participants into the study.
  This study which includes three research sites will be taken as preliminary strata via the simple random sampling technique. Lottery method as one of the oldest and commonly used approach would then be followed to recruit the sample size. Screening of the participants would be taken place in the first round based on the inclusion and exclusion criteria. The eligible participants would be assigned with a code in the second round before recruiting the participant into the study. Lottery method (law of chance) would then be follow to allocate the participants randomly into treatment or control groups in the study sites.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): A total of 30 participants would be exposed to the nursing care training (intervention) randomly.
  Interventions: Behavioral: Transitional Care Training Program
- Control Group (No Intervention): A sample of 30 study participants would not be exposed to the training and would be kept in the control group. They would be a group who would receive usual care and routine awareness by their health care professionals.

INTERVENTIONS:
Behavioral: Transitional Care Training Program — A nursing based transitional care training intervention would be carried out to prepare the family caregivers to take care of their elderly stroke survivors at home. The intervention would be carried out for a tentative time of 2 to 3 hours to educate the family caregivers at their homes after hospitalization. The study participants would be evaluated after 8 weeks of the intervention. A structured, validated and literature based assessment checklist will be devised to assess the usefulness and feasibility of the intervention. Assistance of senior nurses and health professionals, specialized in stroke care will be taken during the training part of the program.
  Arms: Intervention Group

SUMMARY:
The main intention of the study is to understand the need and feasibility of transitional care training program among family caregivers of geriatric stroke survivors in Pakistan

DETAILED DESCRIPTION:
The purpose of the study is to explore the training needs of family caregivers of caring their elderly stroke patients at homes in Pakistan. Secondly the study aims to develop transitional care training program based on the identified needs for family caregivers of geriatric stroke survivors. Furthermore; the study intends to evaluate the feasibility/efficacy of transitional care training program among family caregivers of geriatric stroke survivors.

ELIGIBILITY:
Inclusion Criteria:

* Family caregivers of both genders geriatric stroke survivors will be included
* Family caregivers who care patients both with the Ischemic/hemorrhagic stroke
* Caregivers who have taken care of the patient at least with 1-time hospitalization
* Family caregivers who have taken care for at least 1-weeks at home.

Exclusion Criteria:

* Family Caregivers who are not willing to participate in the study
* Caregivers who has taken with any training regarding the stroke transitional care

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Physical care measured via Training Evaluation Assessment Checklist (TEAC) Questionnaire | Upto 7 months
  Physical care of the geriatric population having a stroke will be evaluated using the physical care section of the standardized Training evaluation assessment checklist (TEAC) questionnaire developed from the qualitative work package of the protocol. This part of the questionnaire includes Hygiene care, range of motion, Bedsore prevention, falls prevention, medication administration, dietary care and elimination care etc. The mean scores will be calculated for the overall population to find the effectiveness of the training program for the geriatric stroke population as compared to the control group.
Psychological care measured via Training Evaluation Assessment Checklist (TEAC) Questionnaire | Upto 7 months
  Psychological care of the geriatric with stroke will be assessed using a psychological section of the standardized Training Evaluation Assessment Checklist (TEAC) questionnaire developed from the qualitative work package of the protocol. This part of the questionnaire includes evaluation of the psychological needs and stress management activities. The mean scores will be calculated for the overall population to find the effectiveness of the training program for the geriatric stroke population as compared to the control group.
Social Care measured via Training Evaluation Assessment Checklist (TEAC) | Upto 7 months
  Social care of the geriatric population with stroke will be assessed using a social care section of the standardized Training Evaluation Assessment Checklist (TEAC) questionnaire developed from the qualitative work package of the protocol. In this domain, TEAC questionnaire includes questions related to social care and spiritual care. The mean scores will be calculated for the overall population to find the effectiveness of the training program for the geriatric stroke population as compared to the control group.
Training Need Assessment | Upto 2 months
  To explore the training needs of family caregivers of caring their elderly stroke patients at homes in Pakistan. (Qualitative Exploration). Training needs of the study participants would be explored qualitatively with the study guided questions.
Training Program Development | Upto 2 months
  To develop transitional care training program based on the identified needs for family caregivers of geriatric stroke survivors. (Based on qualitative parameters during need assessment). A nursing based transitional care training intervention would be planned to prepare family care givers of geriatric stroke survivors.

CONTACTS AND LOCATIONS:
Overall Officials: Sardar Ali, PhD Nursing Scholar, Principal Investigator — Khyber Medical University Peshawar; Dildar Muhammad, PHD Nursing, Study Director — Khyber Medical University Peshawar
Locations (3):
- Pakistan (3):
  - MTI- Lady Reading Hospital (LRH), Peshawar, Khyber Pakhtunkhwa
  - MTI-HMC (Medical Teaching Institution-Hayatabad Medical Complex), -Peshawar, Peshawar, Khyber Pakhtunkhwa
  - MTI-KTH (Medical Teaching Institution-Khyber Teaching Hospital), Peshawar-Pakistan, Peshawar, Khyber Pakhtunkhwa

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interested in the stated study area after its proper monitoring. Data or samples shared will be coded, with no PHI included. Prior permission of the investigators, participants and concerned departments will be obtained.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data requests can be submitted starting 12 months after article publication
Access Criteria: Access can be requested by qualified researchers through proper approval of the investigators.

REFERENCES:
- [Background] Cao LL, Tang YF, Xia YQ, Wei JH, Li GR, Mu XM, Jiang CZ, Jin QZ, He M, Cui LJ. A survey of caregiver burden for stroke survivors in non-teaching hospitals in Western China. Medicine (Baltimore). 2022 Dec 16;101(50):e31153. doi: 10.1097/MD.0000000000031153. PMID 36550813
- [Background] Venketasubramanian N, Yoon BW, Pandian J, Navarro JC. Stroke Epidemiology in South, East, and South-East Asia: A Review. J Stroke. 2017 Sep;19(3):286-294. doi: 10.5853/jos.2017.00234. Epub 2017 Sep 29. PMID 29037005
- [Background] Owolabi MO, Thrift AG, Mahal A, Ishida M, Martins S, Johnson WD, Pandian J, Abd-Allah F, Yaria J, Phan HT, Roth G, Gall SL, Beare R, Phan TG, Mikulik R, Akinyemi RO, Norrving B, Brainin M, Feigin VL; Stroke Experts Collaboration Group. Primary stroke prevention worldwide: translating evidence into action. Lancet Public Health. 2022 Jan;7(1):e74-e85. doi: 10.1016/S2468-2667(21)00230-9. Epub 2021 Oct 29. PMID 34756176
- [Background] Katan M, Luft A. Global Burden of Stroke. Semin Neurol. 2018 Apr;38(2):208-211. doi: 10.1055/s-0038-1649503. Epub 2018 May 23. PMID 29791947
- [Background] Lui SK, Nguyen MH. Elderly Stroke Rehabilitation: Overcoming the Complications and Its Associated Challenges. Curr Gerontol Geriatr Res. 2018 Jun 27;2018:9853837. doi: 10.1155/2018/9853837. eCollection 2018. PMID 30050573
- [Background] Caro CC, Costa JD, Da Cruz DMC. Burden and Quality of Life of Family Caregivers of Stroke Patients. Occup Ther Health Care. 2018 Apr;32(2):154-171. doi: 10.1080/07380577.2018.1449046. Epub 2018 Mar 26. PMID 29578827
- [Background] Steigleder T, Kollmar R, Ostgathe C. Palliative Care for Stroke Patients and Their Families: Barriers for Implementation. Front Neurol. 2019 Mar 6;10:164. doi: 10.3389/fneur.2019.00164. eCollection 2019. PMID 30894836
- [Background] Lou S, Carstensen K, Jorgensen CR, Nielsen CP. Stroke patients' and informal carers' experiences with life after stroke: an overview of qualitative systematic reviews. Disabil Rehabil. 2017 Feb;39(3):301-313. doi: 10.3109/09638288.2016.1140836. Epub 2016 Feb 17. PMID 26882958
- [Background] Anwar A, Saleem S, Aamir A, Diwan M. Organization of Stroke Care in Pakistan. Int J Stroke. 2020 Jul;15(5):565-566. doi: 10.1177/1747493019879663. Epub 2019 Sep 30. PMID 31564238
- [Background] Krishnan S, Hay CC, Pappadis MR, Deutsch A, Reistetter TA. Stroke Survivors' Perspectives on Post-Acute Rehabilitation Options, Goals, Satisfaction, and Transition to Home. J Neurol Phys Ther. 2019 Jul;43(3):160-167. doi: 10.1097/NPT.0000000000000281. PMID 31205230
- [Background] Merati-Fashi F, Dalvandi A, Parsa Yekta Z. Stroke Survivors and Their Family Caregivers' Experiences of Health Information Seeking: A Qualitative Study. Int J Community Based Nurs Midwifery. 2022 Oct;10(4):269-278. doi: 10.30476/IJCBNM.2022.94489.1997. PMID 36274666
- [Background] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476